CLINICAL TRIAL: NCT01891461
Title: A Prospective, Randomized Study to Compare the Addition of Granules of Gelatine + Thrombin to Our Standard of Care (SOC) to Control Post Operative Bleeding in Total Knee Replacement
Brief Title: Study to Compare the Addition of Floseal to Our Standard of Care to Control Post Operative Bleeding in TKR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal (Other)
Collaborators: Baxter Healthcare Corporation (Industry)
Responsible Party: Principal Investigator, Dr Julio Fernandes, MD, MSc, MBA, PhD, Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BS12-000835
Record Dates: First submitted 2013-06-25; First posted 2013-07-03 (Estimated); Last update posted 2017-08-09 (Actual); Status verified 2017-08

CONDITIONS: Intraoperative Bleeding; Post-operative Bleeding
Keywords: total knee arthroplasty; post-operative bleeding; floseal
MeSH Terms: conditions — Blood Loss, Surgical | interventions — FloSeal Matrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Floseal (Experimental): Floseal will be administered during the procedure and prior to release of the tourniquet (if used PRN during the cementing procedure (±10 minutes)) and after the cement has cured, it will be applied to cut, exposed bone ends as well as the intra-articular soft tissue by the use of a delivery syringe. Direct manual pressure with a gauze sponge will be applied following its application for 2 minutes, ensuring that it adheres to the bleeding bone surface.
  Preparation of Floseal requires mixing 5,000 US units of package thrombin (bovine-derived) made up to 5 milliliters of saline solution, to the Gelatin Matrix solution. In this study, 2-4 vials (15-20 mls total) will be used.
  Interventions: Drug: Floseal
- standard of care (No Intervention): For patients randomized to the control arm, the surgery will proceed in an otherwise identical fashion (with release of the tourniquet if used PRN during cementing procedure (±10 minutes)) and hemostasis followed by drain insertion and wound closure.

INTERVENTIONS:
Drug: Floseal — Floseal (5 milliliters) will be applied to the exposed bone in the following order: around the margins of the tibia, the femur (anterior surface, intercondylar notch, exposed medial and lateral condyles) and around the un resurfaced portion of the patella. The other syringes (each of 5 milliliters) will then be applied to the supra-patellar synovium and into the medial and lateral gutters of the knee. No Floseal will be applied outside the knee joint capsule.
  Other Names: Hemostatic Matrix
  Arms: Floseal

SUMMARY:
The purpose of this study is to compare Floseal to our standard of care (SOC) to decrease intraoperative and immediate post-operative bleeding.

DETAILED DESCRIPTION:
A prospective randomized single-blind clinical trial will be conducted at the Hôpital du Sacré-Coeur de Montréal and Hôpital Jean-Talon. All patients admitted for total knee arthroplasty (TKA) between January 2012 and September 2013 Outcome variable: Patient receiving Floseal or SOC

Variables under study:

Primary end point:

Need of transfusion post-op (yes/no, how many)

Patient will be transfused if :

Hg < 80 g/L plus if patient is symptomatic: orthostatic hypotension, tachycardia (pulse> 100/min, hypotension (< 90/60), hx : CVA, CAD)

Secondary end point:

1. Efficacy (during hospital stay)

   * Pre-op and post-op Hg (> 100; 80-100; <80)
   * Hemovac blood drainage (ml)
   * Per operative bleeding (ml)
2. Safety (Follow up: 6wks, 6 ms, 12 ms, 24 ms)

   * Post-op complications: infection, pain, oedema, allergic reaction.
   * Functional outcomes: Knee Society Score (KSS), Western Ontario and McMaster Universities questionnaire (WOMAC), International knee documentation committee form (IKDC)

ELIGIBILITY:
Inclusion Criteria:

* All subjects above 18 years old admitted for a TKA between January 2012 and September 2013at Hôpital du Sacré-Coeur de Montréal (HSCM) and Hôpital Jean-Talon (HJT), Montréal, Quebec, Canada.

  * TKA done without the use of a tourniquet except while cementing only (±10 minutes)
  * TKA done with Smith and Nephew "Genesis II" or Zimmer "NexGen" total knee replacement implants

Exclusion Criteria:

* • Prior osteotomy or knee surgery within last 6-8 wks

  * Active, local infection or systemic infection
  * Participation in any other pharmaceutical or clinical investigation
  * Bleeding disorders (Hemophilia A, Hemophilia B, Von Willebrand disease, factor VIII deficiency, Vitamin K deficiency, Thrombocytopenia (platelets < 50 x 109 per litre)
  * Patients with known allergies to materials of bovine origin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2012-01; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Need of transfusion post-op (yes/no, how many) | post op day 1 to 7

CONTACTS AND LOCATIONS:
Overall Officials: Julio C Fernandes, MDMScMBAPhD, Principal Investigator — Centre Integre Universitaire de Sante et Services Sociaux du Nord de l'ile de Montreal
Locations (1):
- Hopital du sacre coeur de montreal, Montreal, Quebec, Canada